CLINICAL TRIAL: NCT06128902
Title: The Effect of Home-Based Monitoring, Counseling and Exercise Training Applied to Individuals With Chronic Obstructive Pulmonary Disease by Tele-Counselling Method on Repeated Hospitalization and Quality of Life of Individuals
Brief Title: The Effect of Home-Based Monitoring, Exercise Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Hanife DURGUN, Dr, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Tele-nursing
Record Dates: First submitted 2023-11-02; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: COPD Patients
MeSH Terms: interventions — Telemedicine; Educational Status

STUDY DESIGN:
Intervention Model Description: Randomized-control
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): COPD patients
  Interventions: Other: tele health
- Control group (No Intervention): COPD patients

INTERVENTIONS:
Other: tele health — home based exercise and telenursing
  Other Names: education
  Arms: intervention group

SUMMARY:
Chronic obstructive pulmonary disease (COPD); From time to time, significant involvement in dusts or gases and abnormal disease outbreaks are observed, which are observed throughout life in the period when the cause has just emerged, interruption of air flow with disruptions in air flow, shortness of breath, increase in the amount of secretion. Directly or indirectly, very high costs are incurred in COPD care and promotion. While mild stages are treated without directed hospitalization, hospitalizations become more frequent as the disease progresses, and the duration of hospitalization in each acute attack increases compared to the next attack. Acute exacerbations of COPD negatively affect the rates of rehospitalization and emergency service admissions, and the living conditions of this condition, whose long-term cause of death and morbidity has not yet been revealed, do not lead to negative aspects. Exercise programs applied in chronic diseases should include stopping their illnesses, increasing sleep during the disease, stopping inflammatory acuteness, and in addition to treatment, the rest of the patients should be normal. It has been stated that it is more effective than home-based hospital system applications in pulmonary regulation, and it has been taken positively from applications compatible with the basic field, as everywhere in the world. In this direction, the effect of home-based monitoring, education and exercise training applied to individuals with COPD via tele-consultancy method on repeated hospitalization and quality of life is revealed.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the research,
* Diagnosed with COPD,
* Able to use a smartphone,
* Oriented and cooperative,
* Does not have a psychiatric disorder that impairs verbal communication, such as schizophrenia or dementia,
* Having no communication problems.

Exclusion Criteria:

* Having alcohol or drug addiction,
* Those with physical disabilities,
* Illiterate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
repeated hospitalizations | They will be questioned about the number of times they were admitted to hospital due to COPD during 12 weeks.
  after randomization and 12 weeks later

SECONDARY OUTCOMES:
Quality of life that COPD patients | Their quality of life will be evaluated with the SF-36 quality of life (Short Form) immediately after randomization and 12 weeks later.
  after randomization and 12 weeks later

CONTACTS AND LOCATIONS:
Locations (1):
- Nejla KOKSAL, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No